CLINICAL TRIAL: NCT04167865
Title: Effects of Exercise Therapy in Addition to Vacuum Bell in Patients With Pectus Carinatum
Brief Title: Effects of Exercise Therapy on Pectus Excavatum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-14/12
Record Dates: First submitted 2019-11-04; First posted 2019-11-19 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Pectus Excavatum
Keywords: Pectus Excavatum; Orthosis; Exercise
MeSH Terms: conditions — Funnel Chest; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): All patients will be instructed to wear the device for 1 hours for 12 weeks after being instructed on how to use the vacuum bell. The patient's relatives will be asked to keep a book in order to monitor their use. Patients who have not used the device for 5 consecutive days will be excluded from the study. The first group will be given awareness training on using one session orthosis and posture correction.
- Exercise Group (Active Comparator): In addition to the applications to the control group, mobilization, strengthening, posture and segmental breathing exercises will be given . All of these exercises will be combined with segmental breathing exercises depending on the location of the PE. Exercise therapy will be administered by a physiotherapist with 20 years of experience once a week and will be designed as a home program on the remaining days and will be asked to do 45 minutes twice a day (at least 4 times a week). The patient's relatives will be asked to keep a book to monitor the exercise. Patients who do not perform 5 consecutive exercise sessions will be excluded from the study. All treatments will be given for 12 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Orthosis, mobilization, strengthening, posture and segmental breathing exercises
  Arms: Exercise Group

SUMMARY:
Pectus excavatum (PE); It is an anterior chest wall deformity, characterized by varying degrees of depression of the sternum and costal cartilage, usually occurring at birth or in the first year of life. In the treatment of non-severe PE; vacuum bell orthosis and physiotherapy (especially exercise) is recommended as an alternative to surgery. Although there is no literature or consensus about the role of physiotherapy, it is believed that it plays an important role in preventing or correcting deformities and creating a good cosmetic appearance. Therefore, in this study, the investigators aimed to investigate the effectiveness of exercise therapy in addition to vacuum bell therapy.

DETAILED DESCRIPTION:
Pectus excavatum is a relatively common congenital deformity of the chest wall with an incidence of approximately 1 in every 300 births. They find that they have difficulty keeping up with their peers when playing aerobic sports. Furthermore, these patients, already embarrassed by their deformity, will avoid situations where they have to take their shirt off in front of other children, again contributing to less participation in school and team activities. Some patients may exhibit depression by withdrawing from activities with their peers and a declining quality of schoolwork. Most pectus patients have a typical geriatric or pectus posture that includes thoracic kyphosis, forward sloping shoulders and anterior pelvic tilt. A sedentary lifestyle may aggravate this posture, and the poor posture depresses the sternum even further. For this reason, the authors recommend an aggressive pectus posture exercise and breathing program.

Based on the hypothesis that the chest wall is still bendable during adolescence and that the sternum and costal ribs can be reshaped in a normal position with the external suppressor applied on the deformity, the vacuum bell, an orthosis, has been used in the conservative treatment of PE. It is the center of attention as it is an alternative method to surgery for patients.It is thought that by strengthening muscle strength and tone with exercise training, the severity of chest wall deformities can be reduced or at least prevented from progressing. It is stated that a good cosmetic appearance can be provided by exercise training especially by creating a large muscle mass on the anterior chest wall. In the single case study conducted by Canavan and Cahalin (Canavan and Cahalin, 2000) on the effect of exercise training, after 8 weeks of exercise training, the pectus severity index changed by 60% (50 millimeter decreased from 20 millimeter), and during recreational activities and shoulder pain was not found. Therefore, the investigators aimed to investigate the effectiveness of exercise therapy in addition to vacuum bell therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PE by doctor and indicated for the first time orthotic use
* 10-18 years old,
* Discontented with this deformity

Exclusion Criteria:

* Previous orthosis use
* Severe scoliosis (Cobb angle above 20 degrees)
* Having chronic systemic disease
* Having serious psychiatric illness
* Having complex mixed pectus deformity

Ages: 10 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-01-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
External chest wall measurements | Change from baseline External chest wall measurements at 12 weeks
  External chest wall measurements by chest caliper:
  Thorax-caliper measurement: Pectus severity index (T.I.): (T3/T1) * 100 (%) T1: upper edge of the manubrium, T2: Angulus Ludovici , T3: deepest point of the funnel chest, Pectus excavatum: T.I.: < 110
patient's perception of deformity | Change from baseline patient's perception of deformity at 12 weeks
  patient's perception of deformity (0-10):The subject's self-perception of pectus excavatum was obtained through self-report using a scale from 0 (worst self-perception of pectus excavatum) to 10 (best self-perception of pectus excavatum).
Global Rating of Change Score | Through study completion, an average of 12 weeks
  The responses for the Global Rating of Change Score were "much better (2)"; "slightly better (1)"; "stayed the same (0)";"slightly worse (-1)" or "much worse (-2)"
Anthropometric index | Change from baseline Chest anthropometric measurements at 12 weeks
  The A measurement was defined as the largest anteroposterior diameter at the level of the distal third of the sternum, and the B measurement was the largest depth at the same level. The anthropometric index (AI)14 for PEX was defined as the B measurement divided by the A measurement (AI = B/A).
The modified percent depth | Change from baseline modified percent depth at 12 weeks
  At the level of the deepest sternal depression, the sternum, spinous process (posterior midline), and bilateral maximal anterior chest wall projections were marked with temporary ink. The anterior-posterior measurement (cd) is obtained at the lowest depression of the sternum. At the same posterior location the distance from the posterior midline to the right (ad) and left (bd) maximal anterior chest wall projections are recorded. Modified %depth: (ad-cd)/ad*100

SECONDARY OUTCOMES:
New York Posture Rating Chart for posture assessment | Change from baseline score of New York Posture Rating Chart at 12 weeks
  The scores of the remaining 10 body alignment segments are summed, allowing a range ofoverall score between 0 and 100, with a score of 100 representing ideal posture.
The Nuss Questionnaire modified for Adults (Patient form) | Change from baseline score of The Nuss Questionnaire modified for Adults (Patient form) at 12 weeks
  Disease-specific health-related quality of life assessment tool for patients with pectus. The patient version of the NQ-mA includes 12 items, scored 1 to 4. Possible minimum and maximum scores are 12 and 48 in the patient form; higher scores indicate a better quality of life.
The Nuss Questionnaire modified for Adults (Parent form) | Change from baseline score of The Nuss Questionnaire modified for Adults (Parent form) at 12 weeks
  Disease-specific health-related quality of life assessment tool for patients with parent. The parent version of the NQ-mA includes 11 items, scored 1 to 4. Possible minimum and maximum scores are 11 and 44 in the parent form; higher scores indicate a better quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Acibadem University, Istanbul
  - Acıbadem Mehmet Ali Aydınlar University, Department of Physiotherapy and Rehabilitation, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, Informed Consent Form will be shared with the authors every two months
Supporting Information: Study Protocol, ICF
Time Frame: Every 2 months
Access Criteria: Must be an author

REFERENCES:
- [Background] Akkas Y, Gulay Peri N, Kocer B, Gulbahar G, Baran Aksakal FN. The prevalence of chest wall deformity in Turkish children. Turk J Med Sci. 2018 Dec 12;48(6):1200-1206. doi: 10.3906/sag-1807-180. PMID 30541247
- [Background] Bahadir AT, Kuru P, Afacan C, Ermerak NO, Bostanci K, Yuksel M. Validity and reliability of the Turkish version of the nuss questionnaire modified for adults. Korean J Thorac Cardiovasc Surg. 2015 Apr;48(2):112-9. doi: 10.5090/kjtcs.2015.48.2.112. Epub 2015 Apr 5. PMID 25883894
- [Background] Canavan PK, Cahalin L. Integrated physical therapy intervention for a person with pectus excavatum and bilateral shoulder pain: a single-case study. Arch Phys Med Rehabil. 2008 Nov;89(11):2195-204. doi: 10.1016/j.apmr.2008.04.014. PMID 18996250
- [Background] Ewert F, Syed J, Wagner S, Besendoerfer M, Carbon RT, Schulz-Drost S. Does an external chest wall measurement correlate with a CT-based measurement in patients with chest wall deformities? J Pediatr Surg. 2017 Oct;52(10):1583-1590. doi: 10.1016/j.jpedsurg.2017.04.011. Epub 2017 Apr 27. PMID 28499711
- [Background] Haecker FM. The vacuum bell for conservative treatment of pectus excavatum: the Basle experience. Pediatr Surg Int. 2011 Jun;27(6):623-7. doi: 10.1007/s00383-010-2843-7. PMID 21240610
- [Background] Haecker FM, Sesia S. Non-surgical treatment of pectus excavatum. J Vis Surg. 2016 Mar 23;2:63. doi: 10.21037/jovs.2016.03.14. eCollection 2016. PMID 29078491
- [Background] Jaroszewski D, Notrica D, McMahon L, Steidley DE, Deschamps C. Current management of pectus excavatum: a review and update of therapy and treatment recommendations. J Am Board Fam Med. 2010 Mar-Apr;23(2):230-9. doi: 10.3122/jabfm.2010.02.090234. PMID 20207934
- [Background] Lopez M, Patoir A, Costes F, Varlet F, Barthelemy JC, Tiffet O. Preliminary study of efficacy of cup suction in the correction of typical pectus excavatum. J Pediatr Surg. 2016 Jan;51(1):183-7. doi: 10.1016/j.jpedsurg.2015.10.003. Epub 2015 Oct 22. PMID 26526206
- [Background] Rebeis EB, Campos JR, Fernandez A, Moreira LF, Jatene FB. Anthropometric index for Pectus excavatum. Clinics (Sao Paulo). 2007 Oct;62(5):599-606. doi: 10.1590/s1807-59322007000500011. PMID 17952321
- [Background] Schoenmakers MA, Gulmans VA, Bax NM, Helders PJ. Physiotherapy as an adjuvant to the surgical treatment of anterior chest wall deformities: a necessity? A prospective descriptive study in 21 patients. J Pediatr Surg. 2000 Oct;35(10):1440-3. doi: 10.1053/jpsu.2000.16409. PMID 11051146
- [Background] Snyder CW, Farach SM, Litz CN, Danielson PD, Chandler NM. The modified percent depth: Another step toward quantifying severity of pectus excavatum without cross-sectional imaging. J Pediatr Surg. 2017 Jul;52(7):1098-1101. doi: 10.1016/j.jpedsurg.2017.01.053. Epub 2017 Jan 31. PMID 28189448
- [Derived] Alaca N, Alaca I, Yuksel M. Physiotherapy in addition to vacuum bell therapy in patients with pectus excavatum. Interact Cardiovasc Thorac Surg. 2020 Nov 1;31(5):650-656. doi: 10.1093/icvts/ivaa161. PMID 32960955